CLINICAL TRIAL: NCT01999062
Title: Automated Breast Radiation Therapy Using an MR-Guided Process
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Princess Margaret Hospital, Canada (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UHN REB 12-5181-CE
Record Dates: First submitted 2013-06-11; First posted 2013-12-03 (Estimated); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Breast Cancer
Keywords: Breast RT; Breast radiation therapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- IMRT + CT + MR scan (Experimental)
  Interventions: Other: IMRT + CT + MR scan

INTERVENTIONS:
Other: IMRT + CT + MR scan

SUMMARY:
In the proposed research study, we are investigating the feasibility of integrating automated planning tools to MR images acquired using a novel MR-guided linac, for on-line adaptive radiation treatment. However, these on-line automation tools require further technical refinement and clinical validation. The goal of this research proposal is to develop an on-line MR-guided radiation therapy process for adapting breast IMRT treatment. Such an approach will provide early stage breast cancer patients timely access to high-quality adaptive treatments without exposure to additional ionizing radiation.

ELIGIBILITY:
Inclusion Criteria:

* Patients who will receive standard two-field tangential whole breast radiation therapy with dose prescription of 4240 cGy in 16 fractions, 5000 cGy in 25 fractions or 4000 cGy in 16 fractions.
* Female patients with any stage of breast cancer.
* Patients with prior treatment such as surgery or chemotherapy for any type of cancer.
* Able to provide a written informed consent.
* ≥ 18 years of age.

Exclusion Criteria:

* Patients who will not receive 4240 cGy in 16 fractions, 5000 cGy in 25 fractions, or 4000 cGy in 16 fractions
* Males.
* Patients who received partial breast radiation and not the standard dose.
* Patients who are unable to provide informed consent.
* < 18 years of age.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2013-03 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Time between planning of Radiation treatment and the start of radiotherapy | 3 years
The effect of breathing on the position of the heart and lung in treatment plans | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Robert Dinniwell, M.D., Principal Investigator — Princess Margaret Cancer Centre; Tom Purdie, Physicist, Principal Investigator — Princess Margaret Cancer Centre
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada